CLINICAL TRIAL: NCT04538885
Title: Mesenchymal Stem Cell-derived Pleiotropic Factor in Treating Poorly Healed Wounds of Postoperative Incision
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Gansu Provincial Maternal and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-MP-04
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: MSCs-PFs in Treating Poorly Healed Wounds of Postoperative Incision

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No intervention
- experimental group (Experimental): The pleiotropic factor derived from mesenchymal stem cells was smeared on the wound with a dosage of (2.5mg/2cm2)
  Interventions: Biological: The pleiotropic factor derived from mesenchymal stem cells

INTERVENTIONS:
Biological: The pleiotropic factor derived from mesenchymal stem cells — The pleiotropic factor derived from mesenchymal stem cells was smeared on the wound with a dosage of (2.5mg/2cm2), and then the wound was covered with a foam dressing; the dressing was changed every 3 days to reach clinical healing as the end of the trial.
  Arms: experimental group

SUMMARY:
Poor incision healing is a common complication after abdominal surgery, mainly manifested as incision dehiscence, subcutaneous fat liquefaction, malnutrition, and incision infection. Poor healing of the incision will increase the patient's pain and prolong the patient's hospital stay, and the choice of wound treatment is closely related to the wound healing effect. Mesenchymal stem cells mainly rely on paracrine effects to exert their therapeutic effects and obtain better therapeutic effects in wound healing. Here, the pleiotropic factors secreted from mesenchymal stem cells (MSCs-PFs) will be used to treat patients with poor healing after surgery to evaluate its effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Wound size <10X10cm2, the wound base only involves subcutaneous and muscle tissue；
2. Underwent surgical treatment, all incisions were type I, and the incisions healed poorly and delayed healing after 1 week；
3. There is inflammatory reaction at the incision, but no clear indication of infection, or severe infection of the incision.After debridement and dressing change, the infection is controlled and the fresh granulation period is entered
4. Men or women older than 17 years old and younger than 75 years old;
5. Psychologically stable, able to complete the test process.

Exclusion Criteria:

1. Wound size>10X10cm2, the wound base is as deep as the chest and abdominal cavity, causing infection or osteomyelitis in the chest and abdominal cavity;
2. Surgical incision with purulent infection, local purulent secretions can be seen;
3. Those with obvious body temperature and white blood cell elevation, local purulent secretions have positive bacterial culture;
4. Patients with diabetes;
5. Glucocorticoid users;
6. Patients with immune dermatosis;
7. Neoplastic wounds, such as wounds after skin cancer resection, or skin wounds caused by tumor invasion;
8. Psycho-psychological disorders and poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-10 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing time and healing rate | 1 month
  Judgment criteria for incision recovery (4 weeks after treatment): Cure: the patient's incision is completely or basically healed, and the surrounding skin returns to normal; markedly effective: the patient's incision is recovered> 1/2, and the surrounding skin returns to normal; effective: the patient's incision is recovered <1 /2, and the surrounding skin returned to normal; invalid: the patient's incision had no obvious changes, and the surrounding skin color had no obvious improvement.

IPD SHARING:
Plan to Share IPD: Undecided
If any researcher needs it, you can apply to us